CLINICAL TRIAL: NCT06501261
Title: Preliminary Efficacy and Acceptability of CALM Psychotherapy in Chile
Brief Title: CALM Psychotherapy in Patients With Metastatic Cancer in Chile
Acronym: CALM-Ch
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Arturo Lopez Perez (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FALP 001-2022
Record Dates: First submitted 2023-01-17; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Cancer
Keywords: psychotherapy; palliative care
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CALM arm (Experimental): patients receiving CALM sessions
  Interventions: Behavioral: CALM psychotherapy

INTERVENTIONS:
Behavioral: CALM psychotherapy — psychotherapy sessions

SUMMARY:
Patients with metastatic cancer experience multidimensional challenges that increase the risk of emotional distress, which must be addressed by the health team. Chile lacks evidence on effective therapeutic interventions in this population. CALM is a brief, individual (with the presence of a caregiver in one or more sessions) and evidence-based psychotherapy developed at The Princess Margaret Cancer Center. It consists of an intervention of 3 to 6 psychotherapy sessions over a period of 3 to 6 months. The Global CALM program aims to expand CALM research around the world, a program to which FALP has subscribed. Objective: To evaluate the preliminary efficacy of CALM in a sample of patients with metastatic cancer in Chile.

Phase 2 study of preliminary, pseudo-experimental efficacy, without a control group. The study will be carried out in Falp and Corporación Valientes.

DETAILED DESCRIPTION:
Patients with metastatic cancer experience multidimensional challenges that increase the risk of emotional distress, which must be addressed by the health team. Chile lacks evidence on effective therapeutic interventions in this population. CALM is a brief, individual (with the presence of a caregiver in one or more sessions) and evidence-based psychotherapy developed at The Princess Margaret Cancer Center. It consists of an intervention of 3 to 6 psychotherapy sessions over a period of 3 to 6 months. The Global CALM program aims to expand CALM research around the world, a program to which FALP has subscribed. Objective: To evaluate the preliminary efficacy of CALM in a sample of patients with metastatic cancer in Chile.

Phase 2 study of preliminary, pseudo-experimental efficacy, without a control group. The study will be carried out in Falp and Corporación Valientes.

Sample size 34 participants. Sessions will be online, 45 to 50 minutes long. Sessions can be recorded for supervision and training purposes.

ELIGIBILITY:
Inclusion Criteria:

* be ≥18 years of age;
* be fluent in Spanish;
* be able to give informed consent; and
* have received a diagnosis of advanced or metastatic solid tumor cancer with a reduced life expectancy but greater than six months.

Exclusion Criteria:

* significant verbal communication difficulties;
* cognitive impairment indicated by the clinical team or in the patient's file.
* Patients currently in psychotherapy.
* Active suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
depressive symptoms | 3 months
  Patient Health Questionnaire 9- Higher score means higher depression
depressive symptoms | 6 months
  Patient Health Questionnaire 9- Higher score means higher depression
Death anxiety | 3 months
  Death and Dying Distress Scale- Higher score means higher depression
Death anxiety | 6 months
  Death and Dying Distress Scale- Higher score means higher depression

CONTACTS AND LOCATIONS:
Overall Officials: Loreto Fernandez-Gonzalez, Principal Investigator — Fundacion Arturo Lopez Perez
Locations (1):
- Fundacion Arturo Lopez Perez, Providencia, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Supervision Meetings. CALM therapists (IP, co-IP) and the co-investigator team will attend in-person or online supervision meetings offered periodically by GIPPEC and the local research team. To ensure the quality of therapy, compliance with the CALM treatment manual, and delivery of best practices (especially in a diseased population), it is vital that therapists submit audio or video recorded session excerpts. Since CALM developers are located in Toronto, Canada, case discussions and audio or video presentation will be done through online platforms (Teams or Google Meet). These online platforms use secure protocols and are already in use at GIPPEC with other Global CALM participating centers. The videos will not be stored on online platforms. The identification data of the participating patients will not be disseminated in this instance, using only the study ID.
Time Frame: Session recordings will become available during scheduled supervision meetings and will only be watched once.
Access Criteria: GIPPEC faculty and team members